CLINICAL TRIAL: NCT00665262
Title: The Effect of the Combined Use of Naloxone and Tramacet on Postoperative Analgesia in Elderly Patients Having Joint Replacement Surgery: a Prospective Feasibility Study
Brief Title: The Effect of the Combined Use of Naloxone and Tramacet on Postoperative Analgesia in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-06-159; 12177 (Other: REB)
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Arthroplasty
Keywords: analgesia; hip arthroplasty; knee arthroplasty
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): comibined use of tramacet and naloxone infusion perioperatively
  Interventions: Drug: tramacet

INTERVENTIONS:
Drug: tramacet — 2 tablets every 6 hours for 5 days

SUMMARY:
Ten patients 70 years and older having elective total hip/knee replacement surgery will be recruited to receive a continuous IV infusion of naloxone and oral tramacet for analgesia. Postoperative analgesia, satisfaction, side effects, need for rescure analgesia, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* aged 70 years or older able to give consent able to communicate in English having elective hip/knee arthroplasty ASA physical status 1-3

Exclusion Criteria:

* allergies to any of the following: naloxone, tramacet, NSAIDs, sulpha, or local anesthesic contraindication to spinal anesthesia contraindication to use of tramacet or celebrex ASA physical status4 chronic opiod use chronic pain syndrome

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2011-08-12 (Actual)

PRIMARY OUTCOMES:
opoid use post knee/hip arthroplasty | post-op period

SECONDARY OUTCOMES:
incidence of visual analogue scale scores greater than 4 | post-op period

CONTACTS AND LOCATIONS:
Overall Officials: Ngozi Imasogie, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada